CLINICAL TRIAL: NCT03897387
Title: A Post-market, Multi-center, Retrospective Study to Identify Clinical Outcomes and Complications Data From Patients Implanted With the Medacta Versafit Cup DM Prosthesis Who Are at Least Two Years Post Surgery
Brief Title: Post Market, Retrospective Study to Evaluate Patients Implanted With Medacta Versafit Cup DM ™️ 2 Years Post-op
Status: Completed | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MUSA-H-VDM-001
Record Dates: First submitted 2019-03-11; First posted 2019-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Hip Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a post-market, retrospective with one prospective visit, multi- center study, designed to assess the clinical outcomes, surgical details including Anterior or Posterior surgical approach, and collect all complication data of Medacta Versafit Cup DM used for primary or revision total hip arthroplasty at minimum two year post- operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 years and above at the time of consent
2. Able to understand the requirements of the study, provide a written informed consent and comply with the study protocol. Written informed consent must be obtained prior to any study procedure. 3 Patients must be willing to comply with the prospective visit schedule.

4. Patient underwent a primary or revision total hip replacement for any etiology (osteoarthritis, avascular necrosis, inflammatory arthritis, post- traumatic arthritis, hip fracture, failed prior procedures, etc.). 5. Patients must have received a Medacta Versafit Cup DM component 6. Patient must have adequate pre-operative and post-operative radiographs 7. Patients must be at minimum 2 year (24 months) post-treatment 8. The operation was performed by the investigator.

Exclusion Criteria:

1. History of alcoholism
2. Currently on chemotherapy or radiation therapy
3. Habitual use of narcotic pain medications prior to surgery or after surgery for reasons other than hip pain
4. History of a metabolic disorder such as Gout affecting the skeletal system other than osteoarthritis or osteoporosis
5. History of chronic pain issues for reasons other than hip pain
6. Women that are pregnant
7. Patients who underwent Total Hip Arthroplasty (THA) using standard polyethylene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to a total of 528 qualified patients who have undergone primary or revision Total Hip Arthroplasty (THA) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Dislocation rate of Medacta Versafit Cup DM | Minimum 2 years post surgery
  Determine radiographic analysis of component position in millimeters
Implant position fixation and wear | Minimum 2 years post surgery
  Determine by radiographic analysis by measuring Radio Lucent lines in millimeters
Limb length | Minimum 2 years post surgery
  Determined by radiographic analysis by measuring in millimeters
Patient Satisfaction and outcome score | Minimum 2 years post surgery
  Determined by the Hip Disability and Osteoarthritis Outcome Score (HOOS) likert scale score

SECONDARY OUTCOMES:
Patient questionnaire Forgotten Joint Score (FJS) | Minimum 2 years post surgery
  Assessment of awareness of the artificial joint in every day life using the FJS
Patient questionnaire Harris Hip Score (HHS) | Minimum 2 years post surgery
  Assessment of the improvement of clinical outcomes following total hip replacement using the Harris Hip Score
Patient questionnaire Likert Scale Score | Minimum 2 years post surgery
  Assessment of patient satisfaction using the Likert Scale
Gait analysis | Minimum 2 years post surgery
  Assessment of patient limp, use of assistive device
Range of Motion | Minimum 2 years post surgery
  Assessment of contracture
Implant survivorship | Minimum 2 years post surgery
  Determine by radiographic analysis of bone fracture, implant fracture
Surgical Approach | Minimum 2 years post surgery
  Chart review to determine anterior or posterior approach
Implant demographics | Minimum 2 years post surgery
  Chart review to determine type of bearing in Versafit DM
Complications | Minimum 2 years post surgery
  Chart review to determine adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Peak Orthopedics, Lone Tree, Colorado
  - Illinois Bone and Joint Institute, Libertyville, Illinois
  - Texas Orthopedics, Austin, Texas